CLINICAL TRIAL: NCT01538329
Title: Impact of Amantadine on L-DOPA-induced Dyskinesia in Early Parkinson's Disease: a Placebo-controlled Randomized Study (the PREMANDYSK Study)
Brief Title: Amantadine and L-DOPA-induced Dyskinesia in Early Parkinson's Disease
Acronym: PREMANDYSK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11 253 01
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Dyskinesia; L-DOPA; Early introduced treatment; Amantadine
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Amantadine; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amantadine (Experimental): Patients with amantadine
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator): Patients with amantadine placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Amantadine — 200mg / day once daily in the morning and at noon - oral administration -
  Other Names: active drug
  Arms: Amantadine
Drug: placebo — 200mg / day once daily in the morning and at noon - oral administration -
  Other Names: placebo of amantadine
  Arms: Placebo

SUMMARY:
Traditionally amantadine is used at the beginning of Parkinson Disease (PD) treatment in the early stages of the disease, as a modest antiparkinsonian symptomatic treatment. This treatment is usually maintained for no more than the first few months of management, before resorting to drugs deemed more effective as dopamine agonists and lévo-DOPA (L-DOPA). A more modern use of the drug is at a more advanced stage of PD when dyskinesia are already established and become disabling for the patients. There is no data between these two extremes of life stages of Parkinsonism. However, the mechanisms of action of amantadine and the pathophysiology of the motor complications induced by L-DOPA, in particular dyskinesia suggest that the early and prolonged use of amantadine in the early years of management, before L-DOPA-induced dyskinesia have already emerged, should have a positive impact on long-term occurrence and fate of these symptoms, possibly through a glutamatergic mechanism of brain plasticity-of the "disease modification" type.

DETAILED DESCRIPTION:
Traditionally amantadine is used at the beginning of Parkinson Disease (PD) treatment in the early stages of the disease, as a modest antiparkinsonian symptomatic treatment. This treatment is usually maintained for no more than the first few months of management, before resorting to drugs deemed more effective as dopamine agonists and lévo-DOPA (L-DOPA). A more modern use of the drug is at a more advanced stage of PD when dyskinesia are already established and become disabling for the patients. There is no data between these two extremes of life stages of Parkinsonism. However, the mechanisms of action of amantadine and the pathophysiology of the motor complications induced by L-DOPA, in particular dyskinesia suggest that the early and prolonged use of amantadine in the early years of management, before L-DOPA-induced dyskinesia have already emerged, should have a positive impact on long-term occurrence and fate of these symptoms, possibly through a glutamatergic mechanism of brain plasticity-of the "disease modification" type.

The primary purpose of this study is to demonstrate that early introduction of treatment with amantadine (200 mg / d) in the early years of therapeutic care, that is to say during the "honeymoon" of levodopa (early phase of disease <3 years of diagnosis <1 year of L-dopa and lack of complications of levodopa therapy) decreases the rate of subjects with abnormal involuntary dyskinetic movements after 18 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age over 35 years,
* Patients having signed an informed consent before any specific study procedures,
* Patients having a health Insurance Coverage (according to local regulatory requirements),
* Patients suffering from idiopathic Parkinson's disease meeting the definition criteria of the UKPD Brain Bank (Gibb and Lees, 1988),
* Parkinson's disease diagnosed for <3 years,
* Patients receiving treatment with L-DOPA from <1year,
* Lack of complications of levodopa therapy
* Patients receiving a stable antiparkinsonian treatment that may involve, in addition to L-DOPA, a dopamine agonist, a monoamine oxidase-B (MAO-B) or a catecholamine O-methyl transferase (COMT) inhibitor, an anti-cholinergic for at least 2 months before enrollment and in whom we presume it will be possible to maintain this treatment unchanged during the study period (except the dose of L-dopa which can be adjusted during the study after the third month of Phase 1).

Exclusion Criteria:

* Atypical parkinsonian syndromes,
* Drug-induced Parkinsonism,
* Juvenile Parkinson,
* Patients with complications of levodopa therapy
* Inability to keep the current stable antiparkinsonian treatment during the study period, apart from L-DOPA,
* Pretreatment with amantadine,
* amantadine counter-indication
* Neuroleptic treatment,
* Patients with dementia, Mini Mental Status (MMS) <26,
* Patient with behavioral disorder, ECMP item ≥ 3
* Female subjects of childbearing potential without effective contraception

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-03-04 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
after 18 months of Phase 1 of the study | after 18 months of follow-up
  Rate of patient with abnormal involuntary dyskinetic movements (as specifically defined in the protocol) after 18 months of Phase 1 of the study (amantadine versus placebo).

SECONDARY OUTCOMES:
abnormal involuntary dyskinetic movements at the end of phase 3 of the study (wash out) | 22 months after inclusion
  Rate of patients with abnormal involuntary dyskinetic movements at the end of phase 3 of the study (wash out)
motor fluctuations after 18 months of Phase 1 of the study | 18 months after inclusion
  Rate of patients with non-motor fluctuations after 18 months of Phase 1 (defined by the specific scale developed by the Marseille team involved in the project)
Time to onset of dyskinesias | each visits
  Time to onset of dyskinesias defined as the study visit at which the investigator answers "yes" for the first time the question "do you think this patient has dyskinesia as defined in Protocol "

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, MD, Principal Investigator — University Hospital, Toulouse
Locations (18):
- France (18):
  - CHG Aix en Provence, Aix-en-Provence
  - CHU de Bordeaux, Bordeaux
  - CH Jean Rougier, Cahors
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - CHU Dupuytren, Limoges
  - Hopital Lyon, Lyon
  - Hopital de la Timone, Marseille
  - CH Montauban, Montauban
  - hopital Saint Eloi, Montpellier
  - CHu de Nantes, Nantes
  - CH de Narbonne, Narbonne
  - Hopital pitié Salpétriére, Paris
  - Hopital Jean Bernard, Poitiers
  - CH Charles Nicolle, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse